CLINICAL TRIAL: NCT00185458
Title: A 60-month Non-comparative Study on Bleeding Profiles With Levonorgestrel Intrauterine System in Transition From Reproductive Age Contraception to Menopause Age Endometrial Protection During Estrogen Replacement Therapy.
Brief Title: Assessment of the Transfer of Using Levonorgestrel Intrauterine System (LNG IUS) as a Contraceptive to Using it as Part of Hormone Replacement Therapy (HRT).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90660; 300400 (Other: Company Internal)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2009-11-19 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Menopause

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LNG IUS (Experimental): Levonorgestrel Intrauterine System (LNG IUS) (initial in vitro release 20 µg/24h) intrauterine for minimum of 9 months and maximum of 60 months - 2 phases: a) Contraception Phase b) Hormone-Replacement Therapy (HRT) Phase. For outcome measures (vaginal bleeding variables), five 90-day Reference Periods were defined, which were used for comparison during statistical analysis: Reference Period -1 in Contraception Phase; Reference Periods 1-4 in HRT Phase. 90-day reference periods for analyzing vaginal bleeding data are defined by World Health Organization (WHO) guideline. Reference Period -1 is the last 90-day reference period that the subject had before starting the HRT. Reference Period 1 covers the first 90-days of the HRT phase, Reference Period 2 covers days 91 to 180, Reference Period 3 days 181 to 270, and Reference Period 4 days 271 to 360 of the HRT phase.
  Interventions: Drug: LNG IUS

INTERVENTIONS:
Drug: LNG IUS — LNG IUS (initial in vitro release 20 µg/24h) intrauterine for minimum of 9 months and maximum of 60 months - 2 phases: a) Contraception Phase b) HRT Phase. For outcome measures (vaginal bleeding variables), five 90-day Reference Periods were defined, which were used for comparison during statistical analysis: Reference Period -1 in Contraception Phase; Reference Periods 1-4 in HRT Phase. 90-day reference periods for analyzing vaginal bleeding data are defined by WHO guideline. Reference Period -1 is the last 90-day reference period that the subject had before starting the HRT. Reference Period 1 covers the first 90-days of the HRT phase, Reference Period 2 covers days 91 to 180, Reference Period 3 days 181 to 270, and Reference Period 4 days 271 to 360 of the HRT phase.

SUMMARY:
The study has been designed to look at the transfer from using LNG IUS for contraception only, in reproductive age to using it for endometrial protection in menopausal age. The main area of interest in the study is the pattern of any vaginal bleeding that occurs.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer HealthCare AG, Germany. Bayer HealthCare AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Women with intact uterus, regular menstrual cycles and no previous or current climacteric symptoms.

Exclusion Criteria:

* Pregnancy or lactation.
* Previous pelvic infections.
* Abnormal bleeding.
* Abnormal uterine cavity.
* Uterine polyps.
* Genital cancer.
* Liver diseases.
* Alcoholism or drug abuse.

Ages: 46 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 394 (Actual)
Dates: Start 2000-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Belgium (2):
  - Ghent
  - Huy
- Finland (2):
  - Espoo
  - Turku
- Netherlands (4):
  - Heerlen
  - Venlo
  - Zaandam
  - Zwijndrecht
- United Kingdom (3):
  - Cambridge, Cambridgeshire
  - Poole, Dorset
  - Newcastle upon Tyne

REFERENCES:
- [Result] Depypere HT, Hillard T, Erkkola R, Lukkari-Lax E, Kunz M, Rautiainen P, Schram JH. A 60-month non-comparative study on bleeding profiles with the levonorgestrel intrauterine system from the late transition period to estrogen supplemented menopause. Eur J Obstet Gynecol Reprod Biol. 2010 Dec;153(2):176-80. doi: 10.1016/j.ejogrb.2010.08.017. PMID 20888118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only the subjects who reached menopause within max. of 4 years of the contraception phase were eligible for the Hormone-Replacement Therapy (HRT) phase. 58 subjects discontinued the study during the contraception phase before starting the HRT, and 168 subjects who started treatment did not reach menopause.
Pre-assignment Details: 489 subjects were screened: 394 subjects started treatment and 95 subjects failed screening. Intent-to-treat (ITT) population included all subjects (N=394) who had the LNG IUS inserted, or for whom the insertion was attempted. 322 subjects without major protocol deviations were included in the Per protocol set (PPS).
Period: Contraception Phase
Arm/Group | LNG IUS
Started | 394
Completed | 336
Not Completed | 58
Not completed — Adverse Event | 37
Not completed — Lost to Follow-up | 10
Not completed — Protocol Violation | 2
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 7
Period: HRT Phase
Arm/Group | LNG IUS
Started | 168 (168 subjects were eligible for the HRT phase out 336 who completed contraception phase.)
Completed | 141
Not Completed | 27
Not completed — Adverse Event | 18
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | LNG IUS
Number analyzed (Participants) | 394
Age Continuous [Mean (Standard Deviation); unit: years] | 47.8 (1.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 394
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Bleeding Days
Description: Measured by using Subject Diaries (Subject Reported Data)
Time Frame: Last 90 days in Contraception Phase and first 360 days in Hormone-Replacement Therapy (HRT) Phase
Population: Intention to treat population (ITT); all subjects with adequate bleeding diary data. Due to dropouts and missing data the number of subjects do not necessarily sum up to 168, the number of subjects of the ITT, who qualified for the HRT phase.
Measure: Median (Inter-Quartile Range); unit: Bleeding days
Groups:
- Reference Period -1 (Contraception Phase): Patient assessment within the last 90-days before starting the HRT
- Reference Period 1 (HRT Phase): Patient assessment within the first 90-days of the HRT phase
- Reference Period 2 (HRT Phase): Patient assessment within day 91 to 180 of the HRT phase
- Reference Period 3 (HRT Phase): Patient assessment within day 181 to 270 of the HRT phase
- Reference Period 4 (HRT Phase): Patient assessment within day 271 to 360 of the HRT phase
Arm/Group | Reference Period -1 (Contraception Phase) | Reference Period 1 (HRT Phase) | Reference Period 2 (HRT Phase) | Reference Period 3 (HRT Phase) | Reference Period 4 (HRT Phase)
Number analyzed (Participants) | 165 | 154 | 151 | 141 | 132
Bleeding days | 0 [0 to 2] | 0 [0 to 1] | 0 [0 to 2] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Reference Period -1 (Contraception Phase) vs Reference Period 1 (HRT Phase); Time effect tested with Friedman's two-way analysis of variance (ANOVA). The null-hypothesis is that the means are equal at the reference period tested; Test type: Superiority or Other; p = 0.128, Friedman's two-way ANOVA

2. Primary Outcome: Number of Spotting Days
Description: Measured by using Subject Diaries (Subject Reported Data)
Time Frame: Last 90 days in Contraception Phase and first 360 days in HRT Phase
Population: ITT; all subjects with adequate bleeding diary data. Due to dropouts and missing data the number of subjects do not necessarily sum up to 168, the number of subjects of the ITT, who qualified for the HRT phase.
Measure: Median (Inter-Quartile Range); unit: Spotting days
Arm/Group | Reference Period -1 (Contraception Phase) | Reference Period 1 (HRT Phase) | Reference Period 2 (HRT Phase) | Reference Period 3 (HRT Phase) | Reference Period 4 (HRT Phase)
Number analyzed (Participants) | 165 | 154 | 151 | 141 | 132
Spotting days | 4 [0 to 11] | 4 [0 to 10] | 2 [0 to 9] | 1 [0 to 5] | 0 [0 to 6]
Statistical Analysis 1: Comparison: Reference Period -1 (Contraception Phase) vs Reference Period 1 (HRT Phase); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.296, Friedman's two-way ANOVA

3. Primary Outcome: Percentage of Participants With Successful Treatment
Description: Definition of successful treatment:
  * Completion of HRT phase, and
  * Both, the number of bleeding days and the number of spotting days during HRT was equal to or less than during contraceptive phase, and
  * The number of bleeding days and the number of spotting days could be calculated for at least 3 out of the first 4 reference periods in HRT
Time Frame: Last 90 days in Contraception Phase and first 360 days in HRT Phase
Population: ITT; all subjects eligible for the HRT
Measure: Number; unit: Percentage of participants with success
Arm/Group | LNG IUS
Number analyzed (Participants) | 168
Percentage of participants with success | 31

4. Secondary Outcome: Assessment of QOL as Measured by Women's Health Questionnaire
Description: Women's Health Questionnaire (Total Score). For the Total score, the minimum is 36 and maximum is 144. A higher score means the distress and dysfunction are less pronounced.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: ITT. Only the subjects that were eligible for the HRT are included. Due to dropouts and missing data the number of subjects do not necessarily sum up to 168, the number of subjects of the ITT, who qualified for the HRT phase.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Last Measurement Before Start of HRT Phase: Patient assessment at the end of contraception phase
- 6 Months After Start of HRT Phase: Patient assessment about day 180 of the HRT phase
- 12 Months After Start of HRT Phase: Patient assessment about day 360 of the HRT phase
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 165 | 148 | 141
score on a scale | 104.1 (17.75) | 114.4 (16.64) | 112.9 (16.32)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; This is a Friedman's two-way analysis of variance (ANOVA) to test the time effect within the treatment group. The null-hypothesis is that the means are equal at the time points tested; Test type: Superiority or Other; p < 0.001, Friedman's two-way ANOVA

5. Secondary Outcome: Continuation Rates
Description: Percentage of subjects continuing in the study at the given time points.
Time Frame: At entry, at 2 years, at 4 years
Population: ITT. Kaplan-Meier estimator given.
Measure: Number; unit: Percentage of participants continuing
Arm/Group | LNG IUS
Number analyzed (Participants) | 394
Percentage of participants continuing
  At Entry | 100.0
  At 2 Years | 72.3
  At 4 Years | 23.6

6. Secondary Outcome: Progestogenic Symptom 1: Headache (as Measured by a Visual Analogue Scale (VAS))
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 168 | 147 | 139
score on a scale | 23.9 (23.98) | 19.1 (22.57) | 18.2 (23.00)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.027, Friedman's two-way ANOVA

7. Secondary Outcome: Progestogenic Symptom 2: Depressive Mood (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 167 | 147 | 139
score on a scale | 22.3 (25.69) | 11.8 (17.31) | 14.6 (22.10)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Friedman's two-way ANOVA

8. Secondary Outcome: Progestogenic Symptom 3: Acne or Greasy Skin (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 168 | 147 | 139
score on a scale | 8.9 (14.02) | 7.3 (15.38) | 7.6 (15.41)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Friedman's two-way ANOVA

9. Secondary Outcome: Progestogenic Symptom 4: Nausea (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 168 | 147 | 139
score on a scale | 7.5 (13.57) | 5.3 (11.96) | 6.7 (15.32)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Friedman's two-way ANOVA

10. Secondary Outcome: Progestogenic Symptom 5: Edema (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 168 | 147 | 139
score on a scale | 15.7 (20.30) | 12.3 (18.93) | 11.7 (17.65)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.054, Friedman's two-way ANOVA

11. Secondary Outcome: Progestogenic Symptom 6: Decreased Libido (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 166 | 144 | 135
score on a scale | 24.9 (26.29) | 15.6 (22.06) | 17.5 (21.13)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Friedman's two-way ANOVA

12. Secondary Outcome: Climacteric Symptom 1: Hot Flushes (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 167 | 147 | 138
score on a scale | 39.9 (30.21) | 9.4 (14.88) | 11.3 (18.65)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Friedman's two-way ANOVA

13. Secondary Outcome: Climacteric Symptom 2: Sweating Episodes (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 167 | 147 | 138
score on a scale | 43.0 (29.40) | 14.0 (19.95) | 17.0 (21.97)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Friedman's two-way ANOVA

14. Secondary Outcome: Climacteric Symptom 3: Vaginal Dryness (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 167 | 147 | 138
score on a scale | 22.8 (27.96) | 13.1 (20.93) | 16.7 (23.00)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Friedman's two-way ANOVA

15. Secondary Outcome: Climacteric Symptom 4: Sleep Problems (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 167 | 147 | 138
score on a scale | 39.4 (29.71) | 17.1 (21.34) | 19.9 (23.93)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Friedman's two-way ANOVA

16. Secondary Outcome: Climacteric Symptom 5: Irritability (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 167 | 147 | 138
score on a scale | 33.1 (27.40) | 17.2 (19.47) | 19.4 (20.26)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Friedman's two-way ANOVA

17. Secondary Outcome: Climacteric Symptom 6: Breast Tension (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 167 | 147 | 138
score on a scale | 15.5 (22.16) | 13.5 (20.39) | 13.0 (19.42)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.175, Friedman's two-way ANOVA

18. Secondary Outcome: Progestogenic Symptom 7: Hair Loss (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 168 | 147 | 139
score on a scale | 10.0 (15.14) | 9.3 (16.69) | 9.0 (13.63)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.062, Friedman's two-way ANOVA

19. Secondary Outcome: Progestogenic Symptom 8: Greasy Hair (as Measured by a VAS)
Description: Higher value means the symptom is more pronounced. Minimum is 0, maximum is 100.
Time Frame: Last measurement before start of HRT phase, 6 months after start of HRT phase, 12 month after start of HRT phase
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Last Measurement Before Start of HRT Phase | 6 Months After Start of HRT Phase | 12 Months After Start of HRT Phase
Number analyzed (Participants) | 168 | 146 | 139
score on a scale | 14.0 (20.60) | 11.5 (18.85) | 11.1 (18.93)
Statistical Analysis 1: Comparison: Last Measurement Before Start of HRT Phase vs 6 Months After Start of HRT Phase vs 12 Months After Start of HRT Phase; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, Friedman's two-way ANOVA

ADVERSE EVENTS:
Time Frame: The data covers the entire treatment period (contraception phase + HRT phase).
Arm/Group | LNG IUS
Serious Adverse Events (participants affected / at risk) | 25/394
Other Adverse Events (participants affected / at risk) | 357/394
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNG IUS (N=394)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Bladder prolapse (Renal and urinary disorders) | 1
Bronchitis (Infections and infestations) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Colpocele (Reproductive system and breast disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Cystocele (Reproductive system and breast disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Jejunectomy (Surgical and medical procedures) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Palpitations (Cardiac disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Pneumonia (Infections and infestations) | 1
Scar excision (Surgical and medical procedures) | 1
Splenectomy (Surgical and medical procedures) | 1
Thyroidectomy (Surgical and medical procedures) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Varicose vein operation (Surgical and medical procedures) | 1
Venous thrombosis limb (Vascular disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LNG IUS (N=394)
Procedural pain (Injury, poisoning and procedural complications) | 117
Headache (Nervous system disorders) | 59
Back pain (Musculoskeletal and connective tissue disorders) | 47
Influenza (Infections and infestations) | 43
Menopausal symptoms (Reproductive system and breast disorders) | 31
Ovarian cyst (Reproductive system and breast disorders) | 31
Smear cervix normal (Investigations) | 31
Abdominal pain (Gastrointestinal disorders) | 30
Night sweats (Skin and subcutaneous tissue disorders) | 29
Vaginal candidiasis (Infections and infestations) | 29
Breast pain (Reproductive system and breast disorders) | 28
Breast tenderness (Reproductive system and breast disorders) | 27
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 27
Cystitis (Infections and infestations) | 26
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26
Nasopharyngitis (Infections and infestations) | 24
Hypertension (Vascular disorders) | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 20
Bronchitis (Infections and infestations) | 20
Depression (Psychiatric disorders) | 19
Genital haemorrhage (Reproductive system and breast disorders) | 19
Sinusitis (Infections and infestations) | 19
Sleep disorder (Psychiatric disorders) | 18
Weight increased (Investigations) | 17
Abdominal pain lower (Gastrointestinal disorders) | 16
Vaginitis bacterial (Infections and infestations) | 15
Fatigue (General disorders) | 14
Hot flush (Vascular disorders) | 14
Vaginal discharge (Reproductive system and breast disorders) | 14
Vaginal infection (Infections and infestations) | 14
Migraine (Nervous system disorders) | 13
Upper respiratory tract infection (Infections and infestations) | 13
Abdominal distension (Gastrointestinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Metrorrhagia (Reproductive system and breast disorders) | 12
Palpitations (Cardiac disorders) | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11
Urinary tract infection (Infections and infestations) | 11
Vulvovaginal mycotic infection (Infections and infestations) | 11
Dizziness (Nervous system disorders) | 10
Cervical polyp (Reproductive system and breast disorders) | 9
Insomnia (Psychiatric disorders) | 9
Nausea (Gastrointestinal disorders) | 9
Acne (Skin and subcutaneous tissue disorders) | 8
Acute sinusitis (Infections and infestations) | 8
Breast cyst (Reproductive system and breast disorders) | 8
Respiratory tract infection (Infections and infestations) | 8
Tooth infection (Infections and infestations) | 8
Vulvovaginal pruritus (Reproductive system and breast disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators agree to allow the sponsor to review any manuscripts and to negotiate the times and forums of their publication.